CLINICAL TRIAL: NCT00475735
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled, Incomplete Block, Two-period, Crossover Clinical Trial to Study the Safety and Efficacy of MK0249, 10 mg, for Adult Patients, Ages 18 to 55, With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: A Study to Test the Safety and Efficacy of MK0249 in Patients With ADHD (0249-018)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0249-018; 2007_519
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — MK-0249; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- MK-0249 (Experimental): Total time in the study will be ~10 weeks.
  Interventions: Drug: MK0249
- Concerta (Active Comparator): Total time in the study will be ~10 weeks.
  Interventions: Drug: Concerta (methylphenidate)
- Placebo (Placebo Comparator): Total time in the study will be ~10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK0249 — MK-0249, 10 mg per day was taken orally daily. If patients were unable to tolerate 10 mg per day, they were allowed to titrate down to 5 mg per day.
  Arms: MK-0249
Drug: Concerta (methylphenidate) — Titration of Concerta began with two 18-mg capsules (36 mg) for 3 consecutive days, followed by three 18-mg capsules (54 mg) for another 3 consecutive days, ending with four 18-mg capsules (72 mg) for the remainder of the treatment period. If patients were unable to tolerate 72 mg per day, they were allowed to titrate down to 54 mg per day. Concerta was taken orally once daily.
  Other Names: CONCERTA®
  Arms: Concerta
Drug: Placebo — For 4 of the 6 treatment sequences, patients had one 4-week treatment period with placebo of MK-0249 (tablets) and placebo of Concerta (capsules). For patients assigned to active treatments of MK-0249 or Concerta, in order to preserve the blind, placebo of the non-active component was provided, ie, if MK was assigned (tablets), then placebo of Concerta (capsules) was also provided. Each patient was to dose with tablets and capsules, either active or placebo. Placebo was taken orally once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of an investigational treatment for Attention Deficit Hyperactivity Disorder (ADHD) when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 55 years of age (inclusive)
* Patient is an adult with a current DSM-IV diagnosis of ADHD of inattentive or combined subtype, as assessed via a structured interview using the ACDS and AISRS
* Females of child-bearing potential must use acceptable methods of birth control during the study and for 1 month post-therapy

Exclusion Criteria:

* Patient has a history of a neurological disorder resulting in ongoing impairment
* Patient has a lifetime history of a psychotic disorder, bipolar disorder, or post-traumatic stress disorder
* Patient has evidence of ongoing depression
* Patient is sensitive or allergic to methylphenidate
* Patient has glaucoma
* Patient has a previous history of narrowing or blockage of the GI tract
* Patient has a history of a sleep disorder (e.g., insomnia, sleep apnea, nightmares, or night terrors) within 6 months prior to screening
* Patient has a history of a cardiovascular disorder within 6 months prior to screening
* Patient has moderate or severe persistent asthma
* Patient has a history of substance abuse or dependence not in sustained full remission for at least one year according to DSM-IV
* Patient has taken part in a research study within the past 30 days of signing informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Herring WJ, Wilens TE, Adler LA, Baranak C, Liu K, Snavely DB, Lines CR, Michelson D. Randomized controlled study of the histamine H3 inverse agonist MK-0249 in adult attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2012 Jul;73(7):e891-8. doi: 10.4088/JCP.11m07178. PMID 22901359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Dosed: 16 AUG 2007; Last Patient Last Treatment: 04 APR 2008. Six U.S. study centers.
Pre-assignment Details: Pre-Treatment consisted of 2 visits: Screening Visit1 & Baseline Randomization Visit2. Patients continuing after Visit1 entered a 1-wk placebo Run-in period. At Visit2, patients were assessed using the protocol eligibility criteria. Then, if deemed eligible, patients were randomized at Visit2 to one of six 2-period cross-over treatment sequences.
Groups:
- MK-0249 Then Placebo: These participants received MK-0249 during Treatment Period 1 and placebo during Treatment Period 2
- Placebo Then MK-0249: These participants received placebo during Treatment Period 1 and MK-0249 during Treatment Period 2
- MK-0249 Then Concerta: These participants received MK-0249 during Treatment Period 1 and Concerta during Treatment Period 2
- Concerta Then MK-0249: These participants received Concerta during Treatment Period 1 and MK-0249 during Treatment Period 2
- Concerta Then Placebo: These participants received Concerta during Treatment Period 1 and placebo during Treatment Period 2
- Placebo Then Concerta: These participants received placebo during Treatment Period 1 and Concerta during Treatment Period 2
Period: Treatment Period 1
Arm/Group | MK-0249 Then Placebo | Placebo Then MK-0249 | MK-0249 Then Concerta | Concerta Then MK-0249 | Concerta Then Placebo | Placebo Then Concerta
Started | 14 | 13 | 7 | 7 | 16 | 15
Completed | 10 | 11 | 7 | 5 | 14 | 12
Not Completed | 4 | 2 | 0 | 2 | 2 | 3
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — DC due to AE but continuing | 0 | 0 | 0 | 1 | 2 | 2
Not completed — DC due to no efficacy but Continuing | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Washout
Arm/Group | MK-0249 Then Placebo | Placebo Then MK-0249 | MK-0249 Then Concerta | Concerta Then MK-0249 | Concerta Then Placebo | Placebo Then Concerta
Started | 10 | 12 (Includes 1 patient that discontinued Treatment Period 1 but continued the Study.) | 7 | 6 (Includes 1 patient that discontinued Treatment Period 1 but continued the Study.) | 16 (Includes 2 patients that discontinued Treatment Period 1 but continued the Study.) | 14 (Includes 2 patients that discontinued Treatment Period 1 but continued the Study.)
Completed | 10 | 10 | 7 | 6 | 16 | 14
Not Completed | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | MK-0249 Then Placebo | Placebo Then MK-0249 | MK-0249 Then Concerta | Concerta Then MK-0249 | Concerta Then Placebo | Placebo Then Concerta
Started | 10 | 10 | 7 | 6 | 16 | 14
Completed | 10 | 9 | 7 | 4 | 15 | 13
Not Completed | 0 | 1 | 0 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0249 Then Placebo | Placebo Then MK-0249 | MK-0249 Then Concerta | Concerta Then MK-0249 | Concerta Then Placebo | Placebo Then Concerta | Total
Number analyzed (Participants) | 14 | 13 | 7 | 7 | 16 | 15 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (9.2) | 36.9 (11.0) | 39.3 (7.5) | 39.0 (12.3) | 39.8 (11.1) | 36.5 (13.3) | 38.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 5 | 3 | 7 | 27
  Male | 8 | 9 | 5 | 2 | 13 | 8 | 45

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Adult Attention Deficit Hyperactivity Disorder Investigator Symptom Rating Scale (AISRS) Total Score After 4 Weeks of Treatment
Description: The AISRS total score consists of 18 items from the original Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) which were derived based on Diagnostic and Statistical Manual-4 (DSM-IV) criteria for ADHD. The ADHD-RS include 9 items that address symptoms of inattention and 9 items that address symptoms of impulsivity and hyperactivity. Each item is rated from 0 to 3. The AISRS total score can range from 0 to 54. A higher score corresponds to a worse severity of ADHD.
Time Frame: after 4 weeks of treatment
Population: Full Analysis Set (FAS): The FAS included all randomized patients who received at least one dose of study medication. Patients with at least one assessment (baseline or post-randomization) were included in the FAS. Missing data were handled using the data as observed (DAO) approach.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Groups:
- MK-0249: MK-0249, 10 mg per day was taken orally daily. If patients were unable to tolerate 10 mg per day, they were allowed to titrate down to 5 mg per day.
- Concerta: Titration of Concerta began with two 18-mg capsules (36 mg) for 3 consecutive days, followed by three 18-mg capsules (54 mg) for another 3 consecutive days, ending with four 18-mg capsules (72 mg) for the remainder of the treatment period. If patients were unable to tolerate 72 mg per day, they were allowed to titrate down to 54 mg per day. Concerta was taken orally once daily.
Arm/Group | MK-0249 | Concerta | Placebo
Number analyzed (Participants) | 29 | 39 | 48
score on scale | -9.8 [-13.5 to -6.0] | -15.3 [-18.7 to -11.8] | -7.6 [-10.5 to -4.7]
Statistical Analysis 1: Comparison: MK-0249 vs Placebo; Test type: Superiority or Other; p = 0.341, Mixed Models Analysis — Since this is a proof of concept study with one primary hypothesis (AISRS total score for MK-0249 vs. placebo), there is no multiplicity adjustment; The terms were tobacco use, prior stimulant use, time, site, period, sequence, treatment, period-by-time, sequence-by-time, and treatment-by-time
Statistical Analysis 2: Comparison: Concerta vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline in the AISRS Inattentive Subscale Score After 4 Weeks of Treatment
Description: The AISRS inattentive subscale score consists of 9 items from the original ADHD-RS which address inattention. Each item is rated from 0 to 3. The AISRS inattentive subscale score can range from 0 to 27. A higher score corresponds to a worse severity of ADHD inattentiveness.
  Data not reported due to failure of primary hypothesis and program termination.
Time Frame: after 4 weeks of treatment
Reporting Status: Not Posted
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale

3. Other Pre Specified Outcome: Baseline AISRS
Description: Baseline values for all treatment groups are equal because
  the constrained longitudinal data analysis (cLDA) model was used
  (Liang and Zeger, 2000, Sankhyā: The Indian Journal of Statistics, Series B 62, 134-148).
Time Frame: Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | MK-0249 | Concerta | Placebo
Number analyzed (Participants) | 29 | 39 | 48
score on scale | 34.6 (2.80) | 34.6 (2.80) | 34.6 (2.80)

4. Secondary Outcome: >/= 30% AISRS Total Score Responder Rate After 4 Weeks of Treatment;
Description: The AISRS total score consists of 18 items from the original ADHD-RS which were derived based on DSM-IV criteria for ADHD. The ADHD-RS include 9 items that address symptoms of inattention and 9 items that address symptoms of impulsivity and hyperactivity. Each item is rated from 0 to 3. The AISRS total score can range from 0 to 54. A higher score corresponds to a worse severity of ADHD.
  Data not reported due to failure of primary hypothesis and program termination.
Time Frame: after 4 weeks of treatment
Reporting Status: Not Posted
Measure: Number; unit: participants

5. Secondary Outcome: >/=1-point Improvement in the CGI-S Score
Description: The Clinical Global Impression - Severity of Illness Scale (CGI-S) is administered by a trained investigator who rates the severity of a patient's illness at the time of assessment, relative to the investigator's past experience with patients who have an ADHD diagnosis. The scores range from 1 to 7. Higher numbers correspond to more severe illness.
  Data not reported due to failure of primary hypothesis and program termination.
Time Frame: 4 weeks of treatment
Reporting Status: Not Posted
Measure: Number; unit: participants

6. Secondary Outcome: Mean Change From Baseline in the AISRS Hyperactive/Impulsive Subscale Score
Description: The Adult Attention Deficit Hyperactivity Disorder Investigator Symptom Rating Scale (AISRS) hyperactive/impulsive subscale score consists of 9 items from the original Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) which address hyperactivity and impulsivity. Each item is rated from 0 to 3. The AISRS hyperactive/impulsive subscale score can range from 0 to 27. A higher score corresponds to a worse severity of ADHD hyperactivity/impulsivity.
  Data not reported due to failure of primary hypothesis and program termination
Time Frame: 4 weeks of treatment
Reporting Status: Not Posted
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale

7. Secondary Outcome: Mean Change From Baseline in the Conners' Adult ADHD Rating Scale - Observer Screening Version (CAARS-O:SV) Total ADHD Symptom Score.
Description: Conners' Adult ADHD Rating Scale - Observer Screening version (CAARS-O: SV) evaluates DSM-IV-oriented inattention, impulsivity and hyperactivity as well as measures of self-concept. It is a 30-item scale administered by a trained investigator or rater with "cue" questions. Each item is scored from 0 to 3 with higher scores corresponding to worse symptoms. The total score can range from 0 to 90.
  Data not reported due to failure of primary hypothesis and program termination.
Time Frame: 4 weeks of treatment
Reporting Status: Not Posted
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale

8. Secondary Outcome: Mean Change From Baseline in the Clinical Global Impressions-severity of Illness Scale(CGI-S) Score
Description: as for outcome 5
Time Frame: 4 weeks of treatment
Reporting Status: Not Posted
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale

ADVERSE EVENTS:
Time Frame: Patients were assessed for AEs from visit 1 Screening through visit 11 End of Week 9
Description: The population for safety analyses was the All Patients as Treated Set (APaTS)
  population. All patients who were randomized and received at least one dose of study medication were included in the safety analyses. A patient's treatment group was determined by his/her actual treatment.
Arm/Group | MK-0249 | Concerta | Placebo
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/44 | 0/54
Other Adverse Events (participants affected / at risk) | 27/37 | 33/44 | 33/54
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MK-0249 (N=37) | Concerta (N=44) | Placebo (N=54)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Mydriasis (Eye disorders) | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 0
Visual disturbance (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2
dry mouth (Gastrointestinal disorders) | 1 | 10 | 1
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3
nausea (Gastrointestinal disorders) | 3 | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
stomach discomfort (Gastrointestinal disorders) | 1 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1
chills (General disorders) | 1 | 0 | 0
energy increased (General disorders) | 0 | 1 | 0
fatigue (General disorders) | 0 | 4 | 3
feeling hot (General disorders) | 1 | 0 | 0
feeling jittery (General disorders) | 0 | 4 | 2
Influenza like illness (General disorders) | 1 | 1 | 1
Irritability (General disorders) | 2 | 3 | 1
pain (General disorders) | 1 | 0 | 1
pyrexia (General disorders) | 3 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2
Viral infection (Infections and infestations) | 1 | 0 | 1
contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0/27 | 0/36 | 1/43
Aspartate aminotransferase increased (Investigations) | 0/27 | 1/36 | 1/43
Blood bilirubin increased (Investigations) | 0/27 | 1/36 | 0/43
Blood creatine phosphokinase increased (Investigations) | 0/27 | 1/36 | 2/43
Blood lactate dehydrogenase increased (Investigations) | 0/27 | 0/36 | 1/43
Blood pressure increased (Investigations) | 3 | 3 | 3
Weight decreased (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 2
Increased appetite (Metabolism and nutrition disorders) | 3 | 3 | 1
Insulin resistance syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 3 | 4 | 8
Lethargy (Nervous system disorders) | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 0 | 2
Agitation (Psychiatric disorders) | 2 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 7 | 1
Bereavement reaction (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 3
Initial insomnia (Psychiatric disorders) | 1 | 3 | 1
Insomnia (Psychiatric disorders) | 12 | 6 | 7
Libido decreased (Psychiatric disorders) | 1 | 1 | 0
Libido increased (Psychiatric disorders) | 0 | 1 | 0
Middle insomnia (Psychiatric disorders) | 3 | 1 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 3 | 0
Nightmare (Psychiatric disorders) | 2 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Tic (Psychiatric disorders) | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1 | 0
Penile size reduced (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
flatulence (Gastrointestinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.